CLINICAL TRIAL: NCT06980922
Title: The Efficacy and Safety of Guilu Erxian Jiao in the Treatment of Intradialytic Hypotension
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 202400179A3C601
Record Dates: First submitted 2025-05-19; First posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-04

CONDITIONS: Intradialytic Hypotension; End-Stage Renal Disease; Hemodialysis
Keywords: Intradialytic Hypotension; Hemodialysis; Traditional Chinese Medicine; Herbal Medicine; Guilu Erxian Jiao; End-Stage Renal Disease; Randomized Controlled Trial; Kidney Disease; Dialysis Complications; Blood Pressure
MeSH Terms: conditions — Kidney Failure, Chronic; Kidney Diseases

STUDY DESIGN:
Intervention Model Description: This is a two-period, two-sequence crossover trial with a 4-week treatment phase and a 4-week washout period. Participants are randomized in a 1:1 ratio to receive either Guilu Erxian Jiao plus usual care followed by usual care alone, or the reverse sequence.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Participants in Group A will receive Guilu Erxian Jiao (GLJ) plus usual care for 4 weeks, followed by a 4-week washout period, then 4 weeks of usual care alone.
  Interventions: Drug: Guilu Erxian Jiao
- Group B (Active Comparator): Participants in Group B will receive usual care alone for 4 weeks, followed by a 4-week washout period, then 4 weeks of Guilu Erxian Jiao (GLJ) plus usual care.
  Interventions: Drug: Guilu Erxian Jiao

INTERVENTIONS:
Drug: Guilu Erxian Jiao — A traditional Chinese herbal formula composed of Testudinis Carapax, Cervi Cornu, Lycii Fructus, and Ginseng Radix, manufactured by Sun Ten Pharmaceutical Co., Ltd. (License No. 016966). Administered orally at 4 grams per day before meals for 4 weeks.
  Other Names: Jipin Guilu Baishen San

SUMMARY:
The goal of this clinical trial is to learn if Guilu Erxian Jiao, a traditional Chinese herbal medicine, can help manage intradialytic hypotension (IDH), a drop in blood pressure that occurs during hemodialysis in adults. The main questions it aims to answer are:

1. Does Guilu Erxian Jiao reduce the frequency and severity of low blood pressure during dialysis?
2. Is Guilu Erxian Jiao safe to use in patients receiving hemodialysis?

Researchers will compare standard care plus Guilu ErXian Jiao to standard care alone to see if Guilu Erxian Jiao improves blood pressure stability during dialysis.

Participants will:

1. Take Guilu Erxian Jiao once daily in addition to standard care, or receive standard care alone, for 4 weeks, then switch treatments after a 4-week washout period (crossover design).
2. Undergo follow-up assessments at weeks 2 and 4 after each treatment phase.
3. Have their blood pressure monitored before, during (hourly), and after each dialysis session.
4. Report dialysis-related symptoms such as dizziness and fatigue.
5. Receive routine laboratory tests and safety monitoring throughout the study.

DETAILED DESCRIPTION:
1. Clinical Background and Study Rationale

   Intradialytic hypotension (IDH) is defined as a decrease in systolic blood pressure of more than 20 mmHg or a drop of more than 10 mmHg in mean arterial pressure during hemodialysis, often accompanied by symptoms such as dizziness, nausea, or cramps. The incidence of IDH among dialysis patients is approximately 5% to 30%. Risk factors include advanced age, diabetes, female sex, and high body mass index. IDH can cause premature termination of dialysis sessions, resulting in decreased uremic toxin clearance and increased long-term mortality and complications. Severe IDH may lead to bowel ischemia, stroke, or myocardial infarction.

   Common management strategies for IDH include adjusting the dialysis rate, lowering dialysate temperature, avoiding eating during dialysis, and strict sodium intake control. In cases of frequent IDH episodes, drugs such as Midodrine or Vasopressin may be used. However, oral Midodrine can cause side effects such as urinary retention, paresthesia, and pruritus. Its long-term safety in dialysis patients is yet to be confirmed.

   According to Traditional Chinese Medicine (TCM), IDH results from spleen and kidney Qi deficiency, requiring tonification of these organs. Guilu Erxian Jiao (GLJ) is a classical formula composed of Testudinis Carapax, Cervi Cornu, Lycii Fructus, and Ginseng Radix, commonly used to treat Qi deficiency and hypotension. Clinical experience suggests potential efficacy in reducing IDH frequency, but large-scale trials are lacking.

   This trial aims to evaluate the efficacy and safety of GLJ in treating IDH in patients undergoing hemodialysis.
2. Study Design and Methods

   This is a randomized, open-label, crossover clinical trial enrolling 34 patients aged over 18 years who receive thrice-weekly hemodialysis for four hours per session and have a history of IDH. Patients are recruited from nephrology and TCM outpatient clinics and the dialysis unit of Keelung Chang Gung Memorial Hospital.

   Participants will be randomized 1:1 into two groups. Randomization will be performed using a computer-generated random sequence. Participants will be assigned to groups according to sealed envelopes that indicate their allocation. Group A receives GLJ plus conventional treatment for four weeks, followed by a four-week washout period, then four weeks of conventional treatment alone. Group B follows the reverse sequence.

   GLJ (Guilu Erxian Jiao) is administered once daily before meals at a dose of 4 grams for four weeks. The preparation used is Jipin Guilu Baishen San produced by Sun Ten Pharmaceutical Co., Ltd. (License number: 016966).

   Data collected include demographic information, medical history, allergy history, family history, medication history, and socioeconomic status. Evaluations include blood pressure measurements before, during, and after dialysis; frequency of IDH episodes; symptoms such as dizziness and fatigue (via VAS score); laboratory parameters (Na, K, Ca, P, BUN, Cr); and adverse events.

   Follow-up evaluations occur at weeks 2 and 4 after each treatment phase. Each assessment takes approximately 30 minutes.
3. Participant Safety, Compensation, and Withdrawal Rights

   Guilu Erxian Jiao is generally well tolerated. Reported side effects in prior studies include mild dry mouth and constipation. During the study, blood and biochemical parameters will be regularly monitored to detect any possible adverse effects.

   If allergic reactions or serious adverse events occur during the trial, the participant will be withdrawn from the study and provided with appropriate medical evaluation and care.

   Participants may voluntarily withdraw from the study at any time without providing a reason and without any impact on their standard medical care. Likewise, the principal investigator reserves the right to terminate a participant's involvement or discontinue the trial at any time for safety or administrative reasons.

   In case of adverse events or injuries resulting from participation in this study, and if they occur in accordance with the approved protocol, the institution and the principal investigator will be legally responsible for providing necessary compensation. However, no compensation will be provided for anticipated side effects explicitly stated in the study protocol. In addition to compensation, the hospital will also provide professional medical care and consultation at no cost for treating the injury.
4. Data Privacy and Confidentiality

   Participant identities will be anonymized using unique study codes, and no personally identifiable information (e.g., name, medical record number) will appear in the case reports or publications. Study data will be securely stored in locked cabinets and password-protected, encrypted folders for at least two years after the end of the study. Only the principal investigator, authorized research team members, auditors, the ethics committee, and regulatory authorities will have access to the original data for monitoring and auditing purposes. The research team is committed to maintaining confidentiality and protecting participants' privacy throughout the study.
5. Statistical Analysis

   Sample size calculation was based on previous studies with a significance level of 0.05 and power of 0.99, resulting in a required 28 participants; with an estimated 20% dropout rate, 34 participants will be enrolled.

   Statistical analyses include Student's t-test, Chi-square test, ANOVA, and paired t-tests as appropriate. Non-parametric tests will be used if data are not normally distributed. All efficacy analyses will be performed using the intention-to-treat (ITT) principle, including all randomized participants who received at least one dose of study intervention. A one-sided alpha of 0.05 defines statistical significance.
6. IRB Review and Approval This study has been reviewed and approved by the Institutional Review Board of Chang Gung Memorial Hospital, Keelung Branch (IRB No. 2402010026, Protocol Version 5, approved on 2025/03/12).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Undergoing maintenance hemodialysis three times per week, 4 hours per session
* History of intradialytic hypotension (IDH)
* Willing and able to provide written informed consent

Exclusion Criteria:

* Pregnant or lactating women
* Severe comorbid illness, such as cancer, stroke, or liver cirrhosis
* Inability to comply with study medication regimen
* Regular use of antihypertensive medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2027-05-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Frequency of Intradialytic Hypotension Episodes | From baseline through the entire 16-week crossover study, including each 4-week treatment phase and follow-up assessments conducted at 2 and 4 weeks after each treatment phase
  Number of intradialytic hypotension (IDH) episodes, defined as a drop in systolic blood pressure >20 mmHg or mean arterial pressure (MAP) >10 mmHg, recorded during each dialysis session.

SECONDARY OUTCOMES:
Change in Blood Pressure Before, During, and After Dialysis | From baseline through the entire 16-week crossover study, including each 4-week treatment phase and follow-up assessments conducted at 2 and 4 weeks after each treatment phase
  Systolic and diastolic blood pressure measurements are collected before dialysis, hourly during dialysis, and after each dialysis session, then averaged for comparison between treatment phases.
Visual Analogue Scale (VAS) Scores for Dialysis-Related Clinical Symptoms | Assessments are conducted after each dialysis session throughout the 16-week crossover study, including each 4-week treatment phase and follow-up assessments at 2 and 4 weeks after each treatment phase, starting from baseline
  Patient-reported dialysis-related clinical symptoms, such as dizziness and fatigue, are measured using a 0-10 Visual Analogue Scale (VAS) at designated time points throughout the study.
Changes in Laboratory Parameters (Na, K, Ca, P, BUN, Cr) | At baseline and at week 4, 8, 12, and 16 of the study
  Serum levels of sodium, potassium, calcium, phosphate, blood urea nitrogen, and creatinine measured at specified time points to assess biochemical changes.
Adverse Events Related to Guilu Erxian Jiao | Throughout the entire 16-week study period
  All adverse events reported by participants, including dry mouth, constipation, and other symptoms, recorded and monitored throughout the study.
Dialysis Nurse Interventions for IDH | During each dialysis session throughout the 16-week crossover study, including each 4-week treatment phase, and follow-up assessments conducted at 2 and 4 weeks after each treatment phase
  Clinical interventions performed by dialysis nurses in response to intradialytic hypotension, including ultrafiltration adjustment, lowering dialysate temperature, and physician-directed interventions such as fluid administration or early termination of dialysis, as well as other standard nursing responses to IDH, will be recorded at each dialysis session during all study phases.

CONTACTS AND LOCATIONS:
Overall Officials: Huan-Hsuan Hsu, M.D., Principal Investigator — Department of Chinese Medicine, Keelung Chang Gung Memorial Hospital
Locations (1):
- Keelung Chang Gung Memorial Hospital, Keelung, Taiwan

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to privacy protection concerns and no current plan for secondary data use.

REFERENCES:
- [Background] Brunelli SM, Cohen DE, Marlowe G, Van Wyck D. The Impact of Midodrine on Outcomes in Patients with Intradialytic Hypotension. Am J Nephrol. 2018;48(5):381-388. doi: 10.1159/000494806. Epub 2018 Nov 13. PMID 30423552
- [Background] Jindal K, Chan CT, Deziel C, Hirsch D, Soroka SD, Tonelli M, Culleton BF; Canadian Society of Nephrology Committee for Clinical Practice Guidelines. Hemodialysis clinical practice guidelines for the Canadian Society of Nephrology. J Am Soc Nephrol. 2006 Mar;17(3 Suppl 1):S1-27. doi: 10.1681/ASN.2005121372. No abstract available. PMID 16497879
- [Background] Flythe JE, Xue H, Lynch KE, Curhan GC, Brunelli SM. Association of mortality risk with various definitions of intradialytic hypotension. J Am Soc Nephrol. 2015 Mar;26(3):724-34. doi: 10.1681/ASN.2014020222. Epub 2014 Sep 30. PMID 25270068
- [Background] Morfin JA, Fluck RJ, Weinhandl ED, Kansal S, McCullough PA, Komenda P. Intensive Hemodialysis and Treatment Complications and Tolerability. Am J Kidney Dis. 2016 Nov;68(5S1):S43-S50. doi: 10.1053/j.ajkd.2016.05.021. PMID 27772642
- [Background] Flythe JE, Inrig JK, Shafi T, Chang TI, Cape K, Dinesh K, Kunaparaju S, Brunelli SM. Association of intradialytic blood pressure variability with increased all-cause and cardiovascular mortality in patients treated with long-term hemodialysis. Am J Kidney Dis. 2013 Jun;61(6):966-74. doi: 10.1053/j.ajkd.2012.12.023. Epub 2013 Mar 6. PMID 23474007
- [Background] Tattersall J, Martin-Malo A, Pedrini L, Basci A, Canaud B, Fouque D, Haage P, Konner K, Kooman J, Pizzarelli F, Tordoir J, Vennegoor M, Wanner C, ter Wee P, Vanholder R. EBPG guideline on dialysis strategies. Nephrol Dial Transplant. 2007 May;22 Suppl 2:ii5-21. doi: 10.1093/ndt/gfm022. No abstract available. PMID 17507427
- [Background] Mo Y, Liu X, Qin X, Huang J, He Z, Lin J, Hu Q, Cai Y, Liu Z, Wang L. Shenfu injection for intradialytic hypotension: a systematic review and meta-analysis. Evid Based Complement Alternat Med. 2014;2014:279853. doi: 10.1155/2014/279853. Epub 2014 Dec 22. PMID 25587340
- [Background] Sands JJ, Usvyat LA, Sullivan T, Segal JH, Zabetakis P, Kotanko P, Maddux FW, Diaz-Buxo JA. Intradialytic hypotension: frequency, sources of variation and correlation with clinical outcome. Hemodial Int. 2014 Apr;18(2):415-22. doi: 10.1111/hdi.12138. Epub 2014 Jan 27. PMID 24467830
- [Background] Kooman J, Basci A, Pizzarelli F, Canaud B, Haage P, Fouque D, Konner K, Martin-Malo A, Pedrini L, Tattersall J, Tordoir J, Vennegoor M, Wanner C, ter Wee P, Vanholder R. EBPG guideline on haemodynamic instability. Nephrol Dial Transplant. 2007 May;22 Suppl 2:ii22-44. doi: 10.1093/ndt/gfm019. No abstract available. PMID 17507425